CLINICAL TRIAL: NCT01938547
Title: Open Label Study to Assess the Efficacy, Safety and Dosing of Clevidipine in Pediatric Patients Undergoing Surgery
Brief Title: Assessment of Efficacy, Safety and Dosing of Clevidipine in Pediatric Participants Undergoing Surgery (PIONEER)
Acronym: PIONEER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDCO-CLV-12-01
Record Dates: First submitted 2013-08-30; First posted 2013-09-10 (Estimated); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Perioperative Blood Pressure Management
Keywords: perioperative; blood pressure; pediatrics; pediatric surgery
MeSH Terms: interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- clevidipine (Experimental): An initial clevidipine IV infusion dose for the adolescent cohort has been specified per protocol. The initial dose for each of the subsequent age cohorts could be modified if necessary, based on the recommendation of the Data and Safety Monitoring Board (DSMB).
  Following the initial dose, clevidipine will be up-titrated every 1.5 minutes, according to participant need, to achieve a systolic blood pressure (SBP) within the pre-specified SBP target range. Doses may be increased by less than doubling, and the time between dose adjustments may be lengthened, as the target blood pressure is approached. The infusion rate may be maintained for up to 96 hours, once the participant's SBP is within the target range, and titrated as necessary to maintain blood pressure within the range.
  Interventions: Drug: clevidipine

INTERVENTIONS:
Drug: clevidipine
  Other Names: Cleviprex; clevidipine butyrate

SUMMARY:
Evaluate the efficacy, safety, and dosing of clevidipine as an intravenous (IV) infusion for blood pressure (BP) management in paediatric participants in the perioperative setting.

DETAILED DESCRIPTION:
This was an open-label study to assess, in a stepwise approach across 4 age cohorts from oldest to youngest (birth to <age 18), the efficacy and safety of clevidipine exposure for a minimum of 30 minutes and up to a maximum of 96 hours in pediatric participants undergoing a surgical procedure with anesthesia for greater than or equal to 1 hour and for whom parenteral IV infusion of antihypertensive therapy for the management of blood pressure was expected.

The reason for initiating clevidipine administration was to keep blood pressure within a pre-specified range during surgery.

After the study completion for Cohort 1 (adolescent patients 12 to less than 18 years), the PIONEER study was placed on partial clinical hold by the FDA; later, the study was terminated by the sponsor. Enrolment of the subsequent cohorts did not take place; results are presented for Cohort 1 only.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age
* Written informed consent obtained before initiation of any study-related procedures
* The enrolling physician determines that the participant will likely require a 15% reduction in BP during the perioperative course
* Intra-arterial line is available for blood pressure monitoring
* Surgical procedure requiring a minimum of 1 hour of anesthesia, in which IV antihypertensive therapy to control BP for at least 30 minutes is anticipated

Exclusion Criteria:

* Administration of an IV or oral antihypertensive agent within 2 hours prior to study drug administration
* Congenital heart disease described as single ventricle
* Evidence of liver failure, severe liver disease, pulmonary disease (e.g. uncontrolled asthma), hyperlipidemia, lipoid nephrosis, lipid dysfunction or acute pancreatitis
* Allergy to soya bean oil or egg lecithin
* Known to be intolerant to calcium channel blockers
* Hemophilia or blood coagulation disorders
* Any serious medical condition which, in the opinion of the investigator, is likely to interfere with study procedures
* Clinically significant abnormal physical findings at the screening evaluation
* Any serious surgical or medical condition which, in the opinion of the investigator, is likely to interfere with study procedures or with the pharmacokinetics or pharmacodynamics of the study drug
* Participant is terminally ill (death likely to occur within 48 hours)
* Use of Methylphenidate, calcium channel blockers, Aripiprazole and other atypical anti- psychotics and antihypertensives used for BP control within 2 hours prior to study drug initiation
* Positive serum or urine pregnancy test for any female of child bearing potential
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment
* Participants who, for any reason, are deemed by the Investigator to be inappropriate for this study
* Participant is a relative of the Investigator or his/her deputy, research assistant, pharmacist, study coordinator, other staff directly involved in the conduct of the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (2):
- United States (2):
  - Stanford Medical Center, Stanford, California
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clevidipine: An initial clevidipine IV infusion dose for the adolescent cohort has been specified per protocol.
  Following the initial dose, clevidipine was up-titrated every 1.5 minutes, according to participant need, to achieve a systolic blood pressure (SBP) within the pre-specified SBP target range. Doses could be increased by less than doubling, and the time between dose adjustments could be lengthened, as the target blood pressure was approached. The infusion rate may have been maintained for up to 96 hours, once the participant's SBP was within the target range, and titrated as necessary to maintain blood pressure within the range.
Period: Overall Study
Arm/Group | Clevidipine
Started | 22
Completed (Overall, 21 patients were treated with study drug; 1 patient was withdrawn prior to treatment start, based on physician's decision.) | 21
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics of the baseline population: male and female adolescent patients (12 to less than 18 years) who required blood pressure management in the perioperative setting.
Groups:
- Clevidipine: An initial clevidipine IV infusion dose for the adolescent cohort has been specified per protocol.
  Following the initial dose, clevidipine will be up-titrated every 1.5 minutes, according to participant need, to achieve a systolic blood pressure (SBP) within the pre-specified SBP target range. Doses may be increased by less than doubling, and the time between dose adjustments may be lengthened, as the target blood pressure is approached. The infusion rate may be maintained for up to 96 hours, once the participant's SBP is within the target range, and titrated as necessary to maintain blood pressure within the range.
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Height [Mean (Standard Deviation); unit: cm] | 158.20 (13.46)
Weight [Mean (Standard Deviation); unit: kg] | 51.49 (13.47)
Baseline Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 111.0 (17.67)
  Diastolic | 63.4 (5.84)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Median Time to Attain the Initial Pre-specified Target SBP Range
Description: Efficacy: Median time to attain the initial pre-specified target SBP range (≥20 mm Hg and ≤ 40 mm Hg apart).
  The reason for initiating clevidipine administration was to keep blood pressure within a pre-specified range during surgery.
  Time to first achieve SBP target range within first 30 minutes. A target systolic blood pressure (SBP) range was specified for each patient prior to study drug initiation and could not be changed for the first 30 minutes of the treatment period. Adolescent patients received an initial weight-based dose of 0.4 μg/kg/minute, to be maintained for the first 1.5 minutes.
  Treatment period: from study drug initiation to termination of infusion (up to 96 hours) was:
  Phase 1: initial dosing (0 to 1.5 minutes); Phase 2: titration and maintenance phase (>1.5 minutes up to 96 hours); Phase 3: transition and termination phase where the study drug is ceased, and the patient is transitioned to an alternative IV or oral antihypertensive if required.
Time Frame: During the first 30 minutes of clevidipine infusion start (baseline).
Population: Safety population: All patients who received any study drug.
Measure: Median (95% Confidence Interval); unit: minutes
Groups:
- Clevidipine: An initial clevidipine IV infusion dose for the adolescent cohort has been specified per protocol.
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
minutes | 7.9 [7.2 to 10.5]

2. Primary Outcome: Efficacy: Number and Percentage of Participants Achieving the Initial Pre-specified Target SBP Range -- During First 30 Min of Clevidipine Infusion
Description: Efficacy: Number and percentage of participants achieving the initial pre-specified target SBP range within first 30 minutes of clevidipine infusion.
Time Frame: During the first 30 minutes of clevidipine infusion start (baseline).
Population: Safety population: All patients who received any study drug. This was the primary population used for the safety analyses.
Measure: Number; unit: participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
participants | 21

3. Primary Outcome: Efficacy: Total Dose to Attain the Initial Pre-specified Target SBP Range
Description: Efficacy: Total dose infused to attain the initial pre-specified target SBP range (≥20 mm Hg and ≤ 40 mm Hg apart) within the first 30 min.
Time Frame: During the first 30 minutes of clevidipine infusion start (baseline).
Population: as for outcome 2
Measure: Median (Full Range); unit: mg
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
mg | 0.28 [0.02 to 0.91]

4. Primary Outcome: Pharmacology: Pharmacodynamic Variable -- Infusion Rate
Description: Pharmacodynamic (PD) variable: infusion rate.
  A target systolic blood pressure (SBP) range was specified for each patient prior to study drug initiation by the Investigator and could not be changed for the first 30 minutes of the treatment period.
  Adolescent patients received an initial weight-based dose of 0.4 μg/kg/minute, to be maintained for the first 1.5 minutes.
Time Frame: Duration of clevidipine infusion (minimum of 30 minutes up to a maximum 96 hours).
Population: as for outcome 2
Measure: Median (Full Range); unit: microgram/kg/min
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
microgram/kg/min | 0.80 [0.4 to 3.2]

5. Primary Outcome: Pharmacology: Clevidipine -- Tmax
Description: Pharmacology: Pharmacokinetic (PK) variables for clevidipine were established by non-compartmental analysis and non-linear mixed effects modelling (NONMEM).
  PK results represent those that were obtained during and after the infusion of clevidipine, started at infusion rate of 0.4 µg/kg/min and then titrated according to the study protocol.
  Tmax: The time it takes for a drug to reach the maximum concentration after administration of a drug.
Time Frame: From 30 minutes before start of infusion up to termination of infusion (minimum of 9 hours up to a maximum of 96 hours).
Population: PK/PD population: All patients who received any study drug, had at least one documented and evaluable blood concentration and/or SBP observation and documented dose records.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
minutes | 51 (47)

6. Primary Outcome: Pharmacology: Clevidipine -- Cmax
Description: Pharmacology: Pharmacokinetic (PK) variables for clevidipine were established by non-compartmental analysis and non-linear mixed effects modelling (NONMEM).
  PK results represent those that were obtained during and after the infusion of clevidipine, started at infusion rate of 0.4 µg/kg/min and then titrated according to the study protocol.
  Cmax: Highest concentration of a drug reached after administration.
Time Frame: From 30 minutes before start of infusion up to termination of infusion (minimum of 9 hours up to a maximum of 96 hours).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
ng/mL | 14.0 (5.6)

7. Primary Outcome: Pharmacology: Clevidipine -- Area Under the Concentration Curve (AUCall)
Description: Pharmacology: Pharmacokinetic (PK) variables for clevidipine were established by non-compartmental analysis and non-linear mixed effects modelling (NONMEM).
  PK results represent those that were obtained during and after the infusion of clevidipine, started at infusion rate of 0.4 µg/kg/min and then titrated according to the study protocol.
  AUC all: Area under the curve, represents the total drug exposure integrated over time.
Time Frame: From 30 minutes before start of infusion up to termination of infusion (minimum of 9 hours up to a maximum of 96 hours).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
min*ng/mL | 1598 (1540)

8. Primary Outcome: Pharmacology: Clevidipine -- Area Under the Concentration Curve Infinity (AUCinf)
Description: Pharmacology: Pharmacokinetic (PK) variables for clevidipine were established by non-compartmental analysis and non-linear mixed effects modelling (NONMEM).
  PK results represent those that were obtained during and after the infusion of clevidipine, started at infusion rate of 0.4 µg/kg/min and then titrated according to the study protocol.
  AUC inf: Area under the curve of the blood concentration from time zero and extrapolated to infinity.
Time Frame: From 30 minutes before start of infusion up to termination of infusion (minimum of 9 hours up to a maximum of 96 hours).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
min*ng/mL | 1598 (1540)

9. Primary Outcome: Pharmacology: Clevidipine -- Volume of Distribution (Vd)
Description: Pharmacology: Pharmacokinetic (PK) variables for clevidipine were established by non-compartmental analysis and non-linear mixed effects modelling (NONMEM).
  PK results represent those that were obtained during and after the infusion of clevidipine, started at infusion rate of 0.4 µg/kg/min and then titrated according to the study protocol.
  Vd: Volume of distribution is defined as the total amount of drug in the body divided by its concentration in plasma.
Time Frame: From 30 minutes before start of infusion up to termination of infusion (minimum of 9 hours up to a maximum of 96 hours).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
mL/kg | 789 (1165)

10. Primary Outcome: Pharmacology: Clevidipine -- Total Clearance (CL)
Description: Pharmacology: Pharmacokinetic (PK) variables for clevidipine were established by non-compartmental analysis and non-linear mixed effects modelling (NONMEM).
  PK results represent those that were obtained during and after the infusion of clevidipine, started at infusion rate of 0.4 µg/kg/min and then titrated according to the study protocol.
  CL: Total Clearance is defined as the rate at which a drug is removed from plasma (mg/min) divided by the concentration of that drug in the plasma (mg/mL).
Time Frame: From 30 minutes before start of infusion up to termination of infusion (minimum of 9 hours up to a maximum of 96 hours).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
mL/min/kg | 113 (54)

11. Primary Outcome: Pharmacology: Clevidipine -- Half-Life (T1/2)
Description: Pharmacology: Pharmacokinetic (PK) variables for clevidipine were established by non-compartmental analysis and non-linear mixed effects modelling (NONMEM).
  PK results represent those that were obtained during and after the infusion of clevidipine, started at infusion rate of 0.4 µg/kg/min and then titrated according to the study protocol.
  T1/2: The half-life of a drug is the time it takes for the amount of a drug's active substance in your body to reduce by half.
Time Frame: From 30 minutes before start of infusion up to termination of infusion (minimum of 9 hours up to a maximum of 96 hours).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
min | 4.3 (3.6)

12. Secondary Outcome: Efficacy: Percent Change in SBP From Baseline at Each Time Point -- During First 30 Min of Infusion Start (Baseline)
Description: Efficacy: Percent Change in SBP From Baseline at Each Time Point -- During First 30 Min of Infusion Start (Baseline).
Time Frame: From infusion start (baseline) to 30 minutes post baseline.
Population: Safety population: All patients who received any study drug.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
percent change from baseline
  1.5 minutes | -0.6 (9.53)
  3.0 minutes: number analyzed (Participants) | 18
  3.0 minutes | -3.4 (8.19)
  4.5 minutes: number analyzed (Participants) | 20
  4.5 minutes | -4.7 (6.68)
  7.5 minutes: number analyzed (Participants) | 20
  7.5 minutes | -11.6 (7.18)
  10.5 minutes | -18.3 (6.89)
  15 minutes | -18.2 (8.09)
  21 minutes: number analyzed (Participants) | 19
  21 minutes | -18.6 (8.28)
  25.5 minutes: number analyzed (Participants) | 19
  25.5 minutes | -19.3 (9.18)
  30 minutes: number analyzed (Participants) | 18
  30 minutes | -20.8 (7.62)

13. Secondary Outcome: Efficacy: Percent Change From Baseline in SBP -- Hourly Measurements -- From 30 Min to 6 Hours of Infusion Start (Baseline)
Description: Efficacy: Percent change from baseline (infusion start) in SBP at each hour after the first 30 minutes of clevidipine infusion up to the cessation of infusion (up to 6 hours from baseline).
Time Frame: At each hour from 30 minutes post-clevidipine infusion start (baseline) to 6 hours from baseline.
Population: Safety population: All patients who received any study drug.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
percent change from baseline
  1 hour: number analyzed (Participants) | 20
  1 hour | -22.9 (9.47)
  1.5 hours: number analyzed (Participants) | 12
  1.5 hours | -18.6 (12.52)
  2 hours: number analyzed (Participants) | 10
  2 hours | -24.1 (11.33)
  3 hours: number analyzed (Participants) | 4
  3 hours | -15.3 (6.47)
  4 hours: number analyzed (Participants) | 4
  4 hours | -21.5 (9.20)
  5 hours: number analyzed (Participants) | 4
  5 hours | -21.4 (14.07)
  6 hours: number analyzed (Participants) | 1
  6 hours | -14.29 (0.0)

14. Secondary Outcome: Efficacy: Percent Change in SBP From Baseline at Each Time Point -- From Cessation of Study Drug Infusion up to 12 Hours
Description: Efficacy: Percent change in SBP from baseline at each time point -- from cessation of study drug infusion and up to 12 hours.
Time Frame: During the first 12 hours (measured at each hour) after cessation of clevidipine infusion.
Population: Safety population: All patients who received any study drug.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
percent change from baseline
  1 hour | -12.2 (22.92)
  2 hours | -12.1 (21.83)
  3 hours: number analyzed (Participants) | 20
  3 hours | -4.9 (25.07)
  4 hours | -2.8 (23.20)
  5 hours: number analyzed (Participants) | 19
  5 hours | -1.1 (21.00)
  6 hours: number analyzed (Participants) | 19
  6 hours | 0.5 (21.76)
  7 hours: number analyzed (Participants) | 18
  7 hours | 1.2 (20.68)
  8 hours: number analyzed (Participants) | 17
  8 hours | -2.7 (20.79)
  9 hours: number analyzed (Participants) | 17
  9 hours | 1.7 (24.21)
  10 hours: number analyzed (Participants) | 17
  10 hours | 0.9 (19.48)
  11 hours: number analyzed (Participants) | 18
  11 hours | -7.1 (18.48)
  12 hours: number analyzed (Participants) | 16
  12 hours | -4.0 (19.83)

15. Secondary Outcome: Efficacy: Number and Percentage of Patients Falling Below the Target Systolic Blood Pressure Range Lower Limit -- During the First 30 Minutes and During the Entire Drug Treatment Period of Clevidipine Infusion
Description: Efficacy: Number and percentage of patients falling below the target systolic blood pressure range lower limit -- during the first 30 minutes and during the entire drug treatment period of clevidipine infusion.
Time Frame: During the first 30 minutes and during the entire drug treatment period (up to a maximum of 96 hours of clevidipine infusion).
Population: Safety population: All patients who received any study drug.
Measure: Number; unit: participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
participants
  First 30 minutes of clevidipine infusion | 1
  Up to 96 hours of clevidipine infusion | 5

16. Secondary Outcome: Efficacy: Number and Percentage of Participants in Whom the SBP Was Within Target Range at Each Hour After the First 30 Minutes of Clevidipine Infusion (up to 6 Hours)
Description: The number and percentage of participants in whom the SBP was within target range at each hour after the first 30 minutes of clevidipine infusion (up to 6 hours).
Time Frame: From 30 minutes after infusion start (baseline) and up to 6 hours post-clevidipine infusion.
Population: Safety population: All patients who received any study drug.
Measure: Number; unit: participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
participants
  SBP within target range at 1 hour | 8
  SBP within target range at 2 hour: number analyzed (Participants) | 12
  SBP within target range at 2 hour | 5
  SBP within target range at 3 hour: number analyzed (Participants) | 6
  SBP within target range at 3 hour | 5
  SBP within target range at 4 hour: number analyzed (Participants) | 4
  SBP within target range at 4 hour | 1
  SBP within target range at 5 hour: number analyzed (Participants) | 4
  SBP within target range at 5 hour | 2
  SBP within target range at 6 hour: number analyzed (Participants) | 1
  SBP within target range at 6 hour | 0

17. Secondary Outcome: Efficacy: Percent Change From Baseline in Heart Rate (HR) -- During First 30 Min of Infusion
Description: Efficacy: Percent change from baseline in heart rate (HR). From infusion start (baseline) to 30 minutes post baseline.
Time Frame: From infusion start (baseline) to 30 minutes post baseline.
Population: Safety population: All patients who received any study drug.
Measure: Mean (Standard Deviation); unit: Percent change in HR from baseline
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
Percent change in HR from baseline
  1.5 minutes | 5.7 (16.89)
  3 minutes: number analyzed (Participants) | 18
  3 minutes | 0.8 (6.80)
  4.5 minutes: number analyzed (Participants) | 20
  4.5 minutes | 0.7 (7.64)
  6 minutes: number analyzed (Participants) | 20
  6 minutes | 2.2 (7.61)
  7.5 minutes: number analyzed (Participants) | 20
  7.5 minutes | 5.4 (10.12)
  9 minutes: number analyzed (Participants) | 19
  9 minutes | 12.2 (17.97)
  10.5 minutes | 10.6 (15.29)
  12 minutes | 11.1 (14.72)
  13.5 minutes: number analyzed (Participants) | 20
  13.5 minutes | 10.7 (14.02)
  15 minutes | 13.7 (19.63)
  16.5 minutes | 14.8 (20.38)
  18 minutes | 12.7 (16.54)
  19.5 minutes: number analyzed (Participants) | 19
  19.5 minutes | 13.0 (14.48)
  21 minutes: number analyzed (Participants) | 19
  21 minutes | 12.2 (13.59)
  22.5 minutes | 14.7 (15.81)
  24.0 minutes: number analyzed (Participants) | 20
  24.0 minutes | 12.9 (13.95)
  25.5 minutes: number analyzed (Participants) | 19
  25.5 minutes | 15.2 (16.26)
  27 minutes: number analyzed (Participants) | 19
  27 minutes | 13.5 (14.10)
  28.5 minutes: number analyzed (Participants) | 18
  28.5 minutes | 14.9 (13.69)
  30 minutes: number analyzed (Participants) | 18
  30 minutes | 13.0 (14.61)

18. Secondary Outcome: Efficacy: Percent Change From Baseline in Heart Rate (HR).
Description: Efficacy: Percent change from baseline in heart rate (HR) -- From 30 Min to 6 Hours From Baseline.
Time Frame: At each hour after 30 minutes post-clevidipine infusion start (baseline) and up to 6 hours.
Population: Safety population: All patients who received any study drug.
Measure: Mean (Standard Deviation); unit: Percent change in HR from baseline
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
Percent change in HR from baseline
  1 hour: number analyzed (Participants) | 20
  1 hour | 11.5 (16.13)
  2 hours: number analyzed (Participants) | 10
  2 hours | 10.68 (12.89)
  3 hours: number analyzed (Participants) | 4
  3 hours | 8.5 (17.64)
  4 hours: number analyzed (Participants) | 4
  4 hours | 13.2 (16.20)
  5 hours: number analyzed (Participants) | 4
  5 hours | 11.3 (12.26)
  6 hours: number analyzed (Participants) | 1
  6 hours | 12.0 (0.00)

19. Secondary Outcome: Efficacy: Percent Change From Baseline in Heart Rate (HR) -- From Cessation of Study Drug Infusion up to 12 Hours
Description: Efficacy: Percent change from baseline in heart rate. At each hour after cessation of clevidipine infusion (up to 12 hours).
Time Frame: At each hour after cessation of clevidipine infusion (up to 12 hours).
Population: Safety population: All patients who received any study drug.
Measure: Mean (Standard Deviation); unit: Percent change in HR from baseline
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
Percent change in HR from baseline
  1 hour | 11.4 (17.03)
  2 hours | 13.2 (17.88)
  3 hours: number analyzed (Participants) | 20
  3 hours | 10.4 (17.30)
  4 hours | 17.0 (29.48)
  5 hours: number analyzed (Participants) | 19
  5 hours | 11.2 (20.83)
  6 hours: number analyzed (Participants) | 19
  6 hours | 12.3 (23.55)
  7 hours: number analyzed (Participants) | 19
  7 hours | 13.48 (22.33)
  8 hours: number analyzed (Participants) | 16
  8 hours | 12.0 (22.71)
  9 hours: number analyzed (Participants) | 19
  9 hours | 19.8 (31.63)
  10 hours: number analyzed (Participants) | 17
  10 hours | 16.8 (24.90)
  11 hours: number analyzed (Participants) | 17
  11 hours | 15.9 (28.31)
  12 hours: number analyzed (Participants) | 16
  12 hours | 13.0 (21.54)

20. Secondary Outcome: Efficacy: Number and Percentage of Participants Requiring Rescue Therapy
Description: Efficacy: Number and percentage of participants who require rescue therapy (i.e. receive any alternative IV antihypertensive drug) at any time during the study drug treatment period.
Time Frame: Minimum of 30 minutes up to a maximum of 96 hours post infusion start (baseline).
Population: Safety population: All patients who received any study drug.
Measure: Number; unit: participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
participants | 0

21. Secondary Outcome: Efficacy: Number and Percentage of Participants Discontinuing Due to Adverse Events
Description: Number and percentage of participants discontinuing the study due to adverse events.
Time Frame: Minimum of 30 minutes up to a maximum of 96 hours post infusion start (baseline).
Population: Safety population: All patients who received any study drug.
Measure: Number; unit: participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 21
participants | 0

ADVERSE EVENTS:
Time Frame: From start of infusion (baseline) to 7 days after the end of clevidipine infusion (minimum of approximately 7.5 days up to a maximum of approximately 11.5 days).
Description: Safety population was used for analysis of safety. Treatment-emergent adverse events (TEAEs) were defined as those adverse events (AEs) occurring after study drug initiation that were either not present at baseline or were present at baseline but increased in severity after study drug initiation.
Groups:
- Clevidipine: An initial clevidipine IV infusion dose for the adolescent cohort as specified per protocol.
Arm/Group | Clevidipine
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clevidipine (N=21)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clevidipine (N=21)
Nausea (Gastrointestinal disorders) | 12 (12)
Constipation (Gastrointestinal disorders) | 10 (10)
Vomiting (Gastrointestinal disorders) | 9 (9)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Sedation (Nervous system disorders) | 2 (2)
Pyrexia (General disorders) | 5 (5)
Fatigue (General disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
After the study completion for Cohort 1 (adolescent patients 12 to less than 18 years), the PIONEER study was put on partial clinical hold by the FDA; later, the study was terminated by the sponsor. Enrolment of the subsequent cohorts did not take place; results are presented for Cohort 1 only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2013-12-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT01938547/Prot_000.pdf
  • Statistical Analysis Plan (2014-05-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT01938547/SAP_001.pdf